CLINICAL TRIAL: NCT02976831
Title: A Phase I Randomized Single-blind Placebo-controlled 2-part Study to Assess the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of AZD0284 Following Single and Multiple Ascending Dose Administration to Healthy Subjects
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of AZD0284 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7800C00001
Record Dates: First submitted 2016-11-09; First posted 2016-11-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Plaque Psoriasis Vulgaris
Keywords: Plaque psoriasis vulgaris
MeSH Terms: interventions — AZD-0284

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD0284 (Experimental): Part 1A:
  Following an overnight fast of at least 10 hours, each subject will receive a single dose of AZD0284 or matching placebo in the form of an oral solution with water. The total volume that the subject will receive (IMP and water) will be 240 mL.
  Part 1B (food cohort):
  Subjects, will receive a single dose of AZD0284 at a dose level in the range of or slightly above the dose level anticipated to yield therapeutic exposure, currently predicted to be achieved with 28 mg AZD0284 at twice daily dosing. The total volume that the subject will receive (IMP and water) will be 240 mL.
  Part 2:
  In Part 2, subjects will receive 1 dose level of AZD0284 (once or twice daily) with water from Day 1 to between (including) Day 7 and Day 14. The total volume that the subject will receive (IMP with water) will be 240 mL. Subjects may be dosed in either the fasted or fed state depending on emerging data from Part 1.
  Interventions: Drug: AZD0284
- Placebo (Active Comparator): Part 1A: Following an overnight fast of at least 10 hours, each subject will receive a single dose of placebo in the form of an oral solution with water. The first cohort will receive 4.0 mg AZD0284 or placebo on Day 1. The actual dose for subsequent cohorts will be determined after review of all available safety or other pertinent data from the previous dose by the SRC Part 1B (food cohort): In Part 1B, subjects, will receive a single dose of placebo at a dose level in the range of or slightly above the dose level anticipated to yield therapeutic exposure, currently predicted to be achieved with 28 mg AZD0284 at twice daily dosing.
  Part 2: In Part 2, each subject will receive 1 dose level of placebo (once or twice daily) with water from Day 1 to between (including) Day 7 and Day 14. The total volume that the subject will receive (placebo with water) will be 240 mL. Subjects may be dosed in either the fasted or fed state depending on emerging data from Part 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0284 — Oral solution, concentration: 2 mg/mL and 15 mg/mL
  Arms: AZD0284
Drug: Placebo — Placebo matching AZD0284 in the form of an oral solution with water.
  Arms: Placebo

SUMMARY:
Plaque psoriasis vulgaris is a chronic inflammatory skin disorder, affecting 1-3% of the population in Europe and the United States of America (USA) and represents one of the most prevalent immune inflammatory diseases. AZD0284 is a potent selective inverse agonist of RORg, which is being developed for the management of psoriasis. The current Phase 1 study investigates the safety, tolerability, food effect, pharmacokinetic (PK) and pharmacodynamic (PD) properties of single and repeated doses of AZD0284. The study will be conducted in healthy subjects. The study will be divided into 2 parts: Part 1 (SAD) and Part 2 (MAD), with Part 1 being split into 2 sub-parts: 1A (fasting) and 1B (fed). The results from this study will form the basis for decisions on future studies. The study will help to identify appropriate, well-tolerated doses that can be administered in subsequent studies in patients with psoriasis.

DETAILED DESCRIPTION:
Plaque psoriasis vulgaris is a chronic inflammatory skin disorder. There are 2 key abnormalities in psoriasis, hyper proliferation of keratinocytes and an inflammatory cell infiltrate, which includes; dendritic cells (DCs), macrophages, natural killer (NK) T cells, mast cells, T cells and neutrophils. There is strong evidence that T cells have an important role in psoriasis, including the fact that T-cell targeted agents are effective in psoriasis therapy. This study is the first time AZD0284 will be given to humans. The current Phase 1 study investigates the safety, tolerability, food effect, pharmacokinetic (PK) and pharmacodynamic (PD) properties of single and repeated doses of AZD0284. The study will be conducted in healthy subjects to avoid interference from disease processes or other drugs. The study will be divided into 2 parts: Part 1 (SAD) and Part 2 (MAD), with Part 1 being split into 2 sub-parts: 1A (fasting) and 1B (fed). The secondary and safety pharmacology of AZD0284 has been investigated using both in vitro and in vivo models. Screening of AZD0284 in a diverse set of in vitro radiolig and binding, enzyme, functional and electrophysiological assays including cardiac ion channels did not identify any off-target activities likely to be relevant in or near the therapeutic exposure range. The inclusion and exclusion criteria are defined such that the selected subjects will be free of any significant illness when included in the study. The selected starting dose for the SAD part (Part 1A) of the study is 4.0 mg AZD0284 (oral solution). The maximum allowed exposure based on the toxicology studies is 127 μmol*h/L (total AUC(0-24,ss)) or 7.35 μmol/L (total Cmax). In Part 1A (SAD study), 6 dose levels and in Part 2 (MAD study), 3 dose levels are planned. In either part, up to 2 additional doses may be added if needed. The results from this study will form the basis for decisions on future studies. The study will help to identify appropriate, well-tolerated doses that can be administered in subsequent studies in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on admission to the Unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria.

   * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the post-menopausal range.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Hormone replacement therapy is not allowed for females to exclude any drug-drug interaction between the hormone replacement therapy and AZD0284

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the PI.
5. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).
6. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

   * Systolic BP (SBP) < 90 mmHg or ≥ 140 mmHg
   * Diastolic BP (DBP) < 50 mmHg or ≥ 90 mmHg
   * Pulse < 45 or > 85 beats per minute (bpm)
7. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12 Lead ECG as considered by the PI that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy. Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.
8. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation)
9. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
10. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g. ventricular hypertrophy or pre-excitation
11. Known or suspected history of drug abuse, as judged by the PI
12. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
13. History of alcohol abuse or excessive intake of alcohol, as judged by the PI.
14. Positive screen for drugs of abuse or cotinine (nicotine) at screening or admission to the Unit or positive screen for alcohol on admission to the Unit prior to the first administration of IMP.
15. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0284.
16. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the PI.
17. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
18. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
19. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening
20. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of investigational product in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.
21. Receipt of live viral or live bacterial vaccines (such as BCG) 3 months prior to randomization on Day 1.
22. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
23. Subjects who have previously received AZD0284
24. Involvement of any Astra Zeneca or study site employee or their close relatives.
25. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
26. Subjects who are vegans or have medical dietary restrictions.
27. Subjects who cannot communicate reliably with the PI.
28. Subject who have increased risk of infection

    * History and/or presence of tuberculosis (TB); positive result for IFN-γ release assay (IGRA) (i.e. QuantiFERON TB-Gold) the test may be repeated if the initial test result is indeterminate. Subjects who have resided in regions where tuberculosis or mycosis are endemic during 90 days before screening or who intend to visit such a region during the duration of the study.
    * Is in a high-risk group for HIV infection within the last 6 months.
    * Subjects with active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
    * Subjects who have received live or attenuated vaccine in the 4 weeks prior to dosing.
    * Subjects with a disease history suggesting abnormal immune function.

    In addition, the following is considered a criterion for the exclusion from the optional genetic component of the study:
29. Previous bone marrow transplant.
30. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) assessed by recording the number of adverse events. | From Screening till Visit 3 (5 to 7 days post final dose)
  Standard adverse event collection. An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) assessed by recording the supine vital signs (BP [supine and standing], pulse and oral body temperature). | From Screening till Visit 3 (5 to 7 days post final dose)
  The following variables will be collected after the subject has rested in the supine position for at least 5 minutes:
  * Systolic BP (mmHg)
  * Diastolic BP (mmHg)
  * Pulse (beats per minute [bpm])
  * Oral body temperature
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) assessed by electrocardiogram (ECG). | From Screening till Visit 3 (5 to 7 days post final dose)
  A 12-lead ECG will be obtained after the subject rested in the supine position for at least 10 minutes (using the sites own ECG machines when not performing dECGs and using the same machine as the dECGs when time points coincide).
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) assessed by digital ECG (dECG) | From Screening till Visit 3 (5 to 7 days post final dose)
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) assessed by telemetry | From Screening till Visit 3 (5 to 7 days post final dose)
Safety and tolerability of AZD0284 following single dosing (Part 1) and multiple ascending oral dosing (Part 2) by physical examination and laboratory assessments (hematology, clinical chemistry and urinalysis). | From Screening till Visit 3 (5 to 7 days post final dose)
  The complete physical examinations will include an assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.

SECONDARY OUTCOMES:
Pharmacokinetics: Observed maximum concentration, taken directly from the individual concentration-time curve (Cmax) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Effect of food on the bioavailability of AZD0284. | From Day 1 till Follow up Visit (5 to 7 days post final dose)
Presence and extent of renal clearance of AZD0284. | Days 1,2, and 3
  The presence and extent of renal clearance of AZD0284 will be assessed by measuring the drug concentrations in urine.
Confirmation of Proof of Mechanism (PoM) of AZD0284. | Screening, Day 1, Day 2 and Day 3
  The Proof of Mechanism (PoM) will be confirmed by demonstrating that oral dosing of AZD0284 reduces IL-17 secretion by ex vivo stimulated whole blood T cells.
Pharmacokinetics: Time to reach maximum concentration, taken directly from the individual concentration-time curve (tmax) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Terminal half-life, estimated as (ln2)/λz (t1/2λz) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUClast) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Area under the plasma concentration-time curve from time zero to t hours after dosing (AUC0-t) of of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Area under the concentration-time curve from time zero extrapolated to infinity. AUC is estimated by AUC(0-last) + Clast/λz where Clast is the last observed quantifiable concentration (AUC) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Apparent volume of distribution for parent drug at steady state, estimated by dividing the Mean Residence Time (MRT) by the apparent clearance (CL/F) (Vss/F) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Apparent volume of distribution for parent drug at terminal phase (extravascular administration), estimated by dividing the apparent clearance (CL/F) by λz (Vz/F) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Apparent clearance for parent drug estimated as dose divided by AUC (CL/F) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: AUC divided by the dose administered (AUC/D) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: AUC0-t divided by the dose administered (AUC0-t/D) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Cmax divided by the dose administered (Cmax/D) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Mean Residence Time (MRT) of AZD0284. | Part 1A and Part 1B: From Day 1 to Day 4 ( at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Ratio of the fed AUC divided by the fasted AUC (Rfed/fasted AUC) of AZD0284. | Part 1B: From Day 1 to Day 4 during Treatment Period 2 (at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose).
Pharmacokinetics: Ratio of the fed Cmax divided by the fasted Cmax (Rfed/fasted Cmax) of AZD0284 | Part 1B: From Day 1 to Day 4 during Treatment Period 2 (at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose)
Pharmacokinetics: Area under the plasma concentration-time curve in the dosing interval (AUCτ) of AZD0284. | Day 1
Pharmacokinetics: AUClast divided by the dose administered (AUClast/D) of AZD0284. | Day 1
Pharmacokinetics: Observed concentration at the end of the dosing interval (Cmin) of AZD0284. | Day 1
Pharmacokinetics: AUCτ divided by the dose administered (AUCτ /D) of AZD0284. | Day 1
Pharmacokinetics: Accumulation ratio for AUCτ estimated by dividing AUCτ from the last dosing day by AUCτ on Day 1 (Rac AUCτ), of AZD0284 | Day 1
Pharmacokinetics: Accumulation ratio for Cmax , estimated by dividing Css,max from the last dosing day by Cmax on Day 1 (Rac Cmax), of AZD0284 | Day 1
Pharmacokinetics: Temporal change, estimated by dividing AUCτ from the last dosing day by AUC on Day 1 (TCP)of AZD0284 | Day 1
Pharmacokinetics: Amount of analyte excreted into the urine from time t1 to t2 (Ae[t1-t2]) of AZD0284 | Day 1
  Urine collection for PK analyses will be performed in Cohort 4.
Pharmacokinetics: Cumulative amount of unchanged drug excreted in urine from time zero to time after dosing (Ae[0-t]) of AZD0284 | Day 1
  Urine collection for PK analyses will be performed in Cohort 4.
Pharmacokinetics: Fraction of dose excreted in urine from time t1 to t2, estimated by dividing Ae(t1-t2) by dose (fe [t1-t2]) of AZD0284 | Day 1
  Urine collection for PK analyses will be performed in Cohort 4.
Pharmacokinetics: Percentage of dose excreted unchanged into the urine from time zero to time t, estimated by dividing Ae(0-t) by dose * 100 (fe[0-t]%)of AZD0284 | Day 1
  Urine collection for PK analyses will be performed in Cohort 4
Pharmacokinetics: Renal clearance (CLR) of AZD0284 | Day 1
  Urine collection for PK analyses will be performed in Cohort 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom